CLINICAL TRIAL: NCT01214473
Title: Prevention of Neonatal Infection in the Indian Community Setting Using Probiotics
Brief Title: Probiotics for Prevention Neonatal Infection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: DSMB stopped the study due to early effectiveness
Sponsor: University of Nebraska (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0332-10 FB; 5R01HD053719 (NIH)
Record Dates: First submitted 2010-09-30; First posted 2010-10-05 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Neonatal Sepsis; Sepsis; Neonatal Infections
Keywords: Clinical sepsis; Pneumonia; Diarrhea; Probiotics; Synbiotics
MeSH Terms: conditions — Neonatal Sepsis; Sepsis; Pneumonia; Diarrhea | interventions — Synbiotics; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic group (Experimental): Once daily oral administration of a probiotic preparation (1 billion cells of Lactobacillus plantarum and 150 mg of fructooligosaccharides) for one week to newborn infants
  Interventions: Dietary Supplement: Synbiotics
- Placebo (Placebo Comparator): Once daily oral administration of maltodextrin for one week to newborn infants
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Synbiotics — Lactobacillus plantarum with fructo-oligosaccharide
  Arms: Probiotic group
Dietary Supplement: Maltodextrin — Only maltodextrin as placebo
  Arms: Placebo

SUMMARY:
Neonatal sepsis (serious infection) continues to be one of the major causes of morbidity and mortality in the newborn period around the world. India, with one of the world's largest populations, continues to struggle with extremely high infant and neonatal mortality rates. Sepsis accounts for 50% of deaths among community born (and 20% of mortality among hospital-born) infants. Closely linked with this is a burgeoning problem of antimicrobial resistance, which is increasingly restricting the therapeutic options for medical care providers. Friendly bacteria called "Probiotics" have been used in multiple infectious and inflammatory disease states in humans. Fructooligosaccharides are sugars found naturally in many fruits and vegetables and also in human breast milk. These sugars reach the colon undigested and serve as food for the friendly bacteria. The current study uses a probiotic preparation containing Lactobacillus plantarum and fructooligosaccharides as an attempt to prevent neonatal infections. Currently no conclusive data are available on the utility of probiotics in such conditions. If successful, such inexpensive preventive therapy can be made available to general public in resource poor countries. Similar preparations can also be used in the western world to prevent similar infectious conditions of the neonatal period, especially in preterm infants where sepsis continues to be a major cause of hospital stay and death.

DETAILED DESCRIPTION:
Our current study is an attempt to put the well known concept of probiotics through rigorous scientific testing before it could be recommended as a prophylactic therapy against neonatal infections. The study will be conducted in India in 8,442 infants who will receive once daily dosing of probiotics for one week. They will be followed for 60 days at home. We have designed the study with enough power to detect a 20% drop in the incidence rate and plan to collect multiple other demographic data from the mothers and infants to help us discern the possible contribution of other confounding risk factors that have been implicated as cofactors in neonatal infection and death.

This will be a randomized controlled clinical trial involving probiotics (Lactobacillus plantarum 10 billion bacteria and 150 mg of fructo-oligosaccharide). We will use our well established three tier monitoring system in the villages. Infants with any adverse event (including sepsis and other infections) will be brought to attached study hospitals for clinical care. Blood and/or CSG culture will be done using Bactec blood culture system and treatment will be provided based on clinical judgment and microbiological analysis of the blood/CSF and/or other findings such as chest X-ray. Data entry will be done on site and transmitted to the principal investigator's institution in the U.S. A data safety monitoring board convened by expert clinicians, neonatologists, and biostatisticians will monitor the study yearly and more frequently if required. Analyzed data will be published in appropriate journals.

ELIGIBILITY:
Inclusion Criteria:

* All newborn infants in the community >24 hours and <72 hours of age
* 2000 g at birth
* Breastfeeding begun by 24 hr of life
* Able to tolerate oral feeds
* Informed consent by parent or guardian

Exclusion Criteria:

* Evidence or suspicion of clinical sepsis before the baby is randomized
* Not on breast feeding by 24 hr
* Inability to establish oral feeds (in case of maternal death or ailment)
* Presence of major congenital anomalies

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4556 (Actual)
Dates: Start 2007-06; Primary Completion 2012-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Clinical sepsis and/or death | During the first 60 days of life
  Incidence of clinical sepsis and/or death

SECONDARY OUTCOMES:
Culture proven sepsis | During the first 60 days of life
  Incidence of culture proven sepsis (Gram-negative vs. Gram-positive)
Other infections | During the first 60 days of life
  Incidence of other infections
Weight gain | During the first 60 days of life
  Weight gained or lost

CONTACTS AND LOCATIONS:
Overall Officials: Pinaki Panigrahi, MD,PhD, Principal Investigator — University of Nebraska
Locations (2):
- India (2):
  - Center for Advanced Research on Alternative Medicine, Bhubaneswar, Odisha
  - Ispat General Hospital, Rourkela, Odisha